CLINICAL TRIAL: NCT03295695
Title: Pilot Study of PET-CT Imaging Using FDG-labeled Human Erythrocytes in Breast Cancer Patient Before and After Neoadjuvant Chemotherapy
Brief Title: PET-CT Imaging Using FDG-labeled Human Erythrocytes in Breast Cancer Patient
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: closure of radiolaboratory
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-19220
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Breast Cancer, Female; Breast Cancer, Male; Breast Neoplasms
Keywords: Chemotherapy induced cardiotoxicity; Tumor blood perfusion
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Fluorodeoxyglucose F18; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cardiac Imaging - All Participants (Experimental): Study agent: 2-deoxy-2-[18F]fluoro-D-glucose (FDG). Fluoro-D-glucose-positron Emission Tomography: Participants will undergo a PET-CT scan with Fluoro-D-glucose-labeled (FDG-labeled) red blood cells (RBCs) within 2 weeks of obtaining an echocardiogram prior to start of chemotherapy. A repeat FDG-RBC PET-CT scan will be completed within two weeks of obtaining their follow-up echocardiogram to determine post-therapy cardiac ejection fraction. If the participant has an echocardiogram obtained prior to completion of chemotherapy, an attempt will be made to obtain a FDG-RBC PET-CT scan within two weeks of the echocardiogram.
  Interventions: Diagnostic Test: Fluoro-D-glucose-positron Emission Tomography; Biological: 2-deoxy-2-[18F]fluoro-D-glucose (FDG); Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: Fluoro-D-glucose-positron Emission Tomography — 2-deoxy-2-[18F]Fluoro-D-glucose-positron Emission Tomography (FDG-PET): within 2 weeks of obtaining first echocardiogram; within two weeks of obtaining follow-up echocardiogram.
  Other Names: FDG-RBC PET-CT scan; Cardiac blood pool imaging
Biological: 2-deoxy-2-[18F]fluoro-D-glucose (FDG) — 2-deoxy-2-[18F]fluoro-D-glucose (FDG) labeled autologous human erythrocytes (RBCs): Approximately 10 mls of packed human erythrocytes are collected from the patient and labeled with ≈5-10 milliCuries of commercially available United States Pharmacopeia (USP)-grade FDG (≈5-10 picograms FDG) (Vendor: Cardinal Health) under sterile conditions in a Good Manufacturing Practice (GMP)-certified laboratory.
  Synthesized RBCs: The cell suspension is manually infused via syringe through an indwelling peripheral venous catheter over the course of 1 minute, using an infusion method approved by the Moffitt Cancer Center (MCC) radiation safety officer.
  Other Names: FDG-labeled RBCs; 18F-fluorodeoxyglucose (FDG)-labeled human erythrocytes
Diagnostic Test: Echocardiogram — Echocardiogram: prior to start of chemotherapy; post-treatment regimen.
  Other Names: Echocardiography

SUMMARY:
This is a single arm, phase 0 study to evaluate the safety and efficacy of PET-CT scans with FDG-labeled RBC in patients with breast cancer.

Cardiac ejection fraction can be calculated and monitored in breast cancer patients during chemotherapy using a FDG-RBC PET-CT scan. The purpose of this study is to determine if calculated cardiac ejection fraction shows high concordance with results from echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed breast cancer and be scheduled for neoadjuvant Trastuzumab- or anthracycline-based chemotherapy.
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >60%).
* Must be able to complete an informed consent process.
* Must have normal organ and marrow function: leukocytes >3,000/μL; absolute neutrophil count >1,500/μL; platelets >100,000/μL; total bilirubin within normal institutional limits; aspartate aminotransferase (AST)[SGOT] / alanine aminotransferase (ALT)[SGPT]: less than 2.5 X institutional upper limit of normal; Creatinine within normal institutional limits - OR - creatinine clearance>60 mL/min/1.73 m^2 for patients with creatinine level above institutional normal.
* Echocardiogram results should be of sufficiently suitable quality (adequate acoustic window access) to provide a reliable ejection fraction range calculation. The cardiac ejection fraction on the pre-treatment echocardiogram should be 50% or higher.
* Participants should be naïve to Trastuzumab or anthracycline chemotherapy prior to enrollment.

Exclusion Criteria:

* Prior history of invasive breast cancer and treatment with anthracycline chemotherapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to FDG.
* Known symptomatic coagulopathies, bleeding diathesis, hemoglobinopathies, or hemolytic anemia.
* Participants should have no clinically significant heart disease such as congestive heart failure. Participants should not have other significant structural heart disease by echocardiogram, or cardiac dysrhythmia on standard of care electrocardiogram that may adversely affect the cardiac imaging results obtained with FDG-RBC PET-CT imaging.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant.
* Found to have a cardiac ejection fraction less than 50% on the pre-treatment echocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac Ejection Fraction (EF) | Up to 12 months
  Calculated cardiac ejection fraction (EF) with a low radiation dose FDG-RBC PET-computed tomography (CT) scan before and after neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Concordance Between FDG-RBC PET-CT and Echocardiogram | Pre-treatment and Post-treatment, up to 12 months
  The concordance will be estimated by the use of Lin's method49 along with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Choi, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/